CLINICAL TRIAL: NCT00258089
Title: A Multicenter, Double-Blind, Randomized Study To Compare The Safety And Efficacy Of Oral Levofloxacin With That Of Ciprofloxacin HCl In The Treatment Of Complicated Urinary Tract Infections In Adults
Brief Title: A Study of the Safety and Effectiveness of Oral Levofloxacin Compared With Oral Ciprofloxacin in the Treatment of Complicated Urinary Tract Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005482
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2010-11

CONDITIONS: Urinary Tract Infections; Bacteriuria; Urologic Diseases; Pyelonephritis; Neurogenic Bladder
Keywords: levofloxacin; urinary tract infections; bacterial infections; bacteriuria; urinary anti-infective agents; urinary infections; quinolones
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria; Urologic Diseases; Pyelonephritis; Urinary Bladder, Neurogenic; Bacterial Infections | interventions — Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin

SUMMARY:
The purpose of the study is to compare the safety and effectiveness of oral levofloxacin (an antibiotic) with that of oral ciprofloxacin in the treatment of complicated urinary tract infections in adults.

DETAILED DESCRIPTION:
Levofloxacin is an antibacterial agent used for the treatment of a many types of acute infections in adults. This is a randomized, double-blind study of the safety and effectiveness of levofloxacin compared with ciprofloxacin in the treatment of adults with a complicated urinary tract infection. Complicated urinary tract infections include those associated with fever, chills, kidney involvement or anatomic and functional abnormalities of the bladder. Patients in one group are treated with 250 mg of levofloxacin taken once daily for 10 days, and the other group is treated with 500 mg of ciprofloxacin, also an antibacterial agent, taken twice daily for 10 days. Patients are followed for 5 to 9 days after completion of treatment (post-therapy) to assess clinical signs and symptoms of infection. Long-term follow up (4 to 6 weeks after the end of treatment) of those patients who respond to therapy provides further evaluation of clinical signs and symptoms. The primary assessments of effectiveness include the microbiological response (the eradication at post-therapy of the infectious organism identified at the start of the study) and the clinical response (the resolution of signs and symptoms at post-therapy compared with those at the start of the study). An additional assessment of efficacy includes the overall clinical response, which is described as cured, improved, or failed. Safety assessments include the incidence of adverse events throughout the study, clinical laboratory tests (hematology, serum chemistry, and urinalysis) and physical examinations at the start of the study and post-therapy. The study hypothesis is that levofloxacin is at least as effective therapeutically and as well tolerated as ciprofloxacin in the treatment of adults with complicated urinary tract infections. Two levofloxacin 125 mg tablets taken orally once daily (and two placebo tablets taken once daily, 12 hours later) for 10 days; or one ciprofloxacin 500 mg tablet and one placebo tablet taken orally twice daily for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a urinary tract infection with complicating factors such as anatomical or functional abnormalities
* capable of taking medication by mouth
* previous antibacterial therapy of less than 24 hours, or previous antibacterial therapy of greater than 24 hours that did not eliminate or stabilize the infection.

Exclusion Criteria:

* Patients having any medical condition that requires antimicrobial therapy to be given intravenously or by hypodermic needle
* complete obstruction of any part of the urinary tract
* inflammation of the prostate gland
* previous allergic or serious adverse reaction to similar antibiotics
* pregnant or nursing females, or those lacking adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 1993-06; Study Completion 1995-01 (Actual)

PRIMARY OUTCOMES:
Clinical response, the resolution of signs and symptoms at post-therapy compared with those at the start of study; Microbiological response, the eradication at post-therapy of infectious organism identified at start of study.

SECONDARY OUTCOMES:
Overall clinical response (described as cured, improved or failed) at long-term follow up; incidence of adverse events throughout the study; change in clinical laboratory tests and physical examinations from start of study to post-therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the safety and effectiveness of oral levofloxacin compared with oral ciprofloxacin in the treatment of complicated urinary tract infections — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=653&filename=CR005482_CSR.pdf